CLINICAL TRIAL: NCT06097780
Title: Phase III Efficacy and Safety of NestaCell® in Moderated Huntington's Disease
Brief Title: Efficacy and Safety of NestaCell® in Huntington's Disease
Acronym: STAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Cellavita Pesquisa Científica Ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAR; U1111-1298-5627 (Other: WHO)
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Huntington Disease
Keywords: STAR; NestaCell ®
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: The trial will evaluate 120 adult patients (male and female) aged 18 to 55 years with Huntington's disease:CAG repeats from 40 to 50; HD diagnostic confidence level (DCL) score of 4;UHDRS Total Functional Capacity (TFC) from 7 to 12, suggesting mild-moderate functional impairment.
  Each patient participates in the trial for approximately 14 months, two months for screening, and twelve months for investigational product administration and follow-up.
Who Masked: Outcomes Assessor
Masking Description: The trial will be two-armed double-blind (participant and investigator's team responsible for outcome assessments).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Arm 1: Nine intravenous placebo administrations in twelve months.
  Interventions: Genetic: NestaCell®
- Intravenous NestaCell® administrations (Experimental): Arm 2: Nine intravenous NestaCell® administrations in twelve months.
  Interventions: Genetic: NestaCell®

INTERVENTIONS:
Genetic: NestaCell® — Human Dental Pulp Stem Cells (hDPSCs).

SUMMARY:
Huntington's disease (HD) is a rare neurodegenerative condition caused by increased CAG trinucleotide repeats in the HTT gene, on chromosome 4. The estimated global prevalence is 2.71 cases per 100,000 inhabitants. In Brazil, it is estimated that 13,000 to 19,000 people carry the gene and 65,000 to 95,000 are descendants at risk.

HD usually manifests itself in the fourth decade of life with motor, cognitive and behavioral symptoms, such as chorea. This condition profoundly affects quality of life and there is no treatment that can modify its course. Tetrabenazine is the only medication approved to control chorea.

A partnership between the Butantan Institute and Cellavita investigates the use of Human Dental Pulp Stem Cells (hDPSCs) to treat HD. NestaCell® was developed, a product based on these cells, which express high levels of BDNF, an important neurotrophic factor for neuronal survival.

Preclinical tests showed that NestaCell® is distributed to several organs, including the central nervous system, being well tolerated in toxicological tests in rats.

In phase I (SAVE) and phase II (ADORE) clinical trials, NestaCell® was administered to patients with HD. The results indicated a significant improvement in motor scores and functional capacity compared to placebo, demonstrating a clinically significant benefit.

NestaCell® also presented a good safety and tolerability profile, with few adverse events related to the product. The results support the conclusion that NestaCell® is safe and well tolerated in HD patients, within the doses tested.

DETAILED DESCRIPTION:
This is a Phase III multicenter, prospective, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of Nestacell® in Huntington's Disease.

After signing the Informed Consent Form (ICF) the patients will perform the V-2 and V-1 screening procedures. In the V-2 the site collects personal data and a physician clinically confirms the HD diagnosis. The patient collects blood for CAG repeats and safety exams. Females with childbearing potential perform a urine pregnancy test. In the V-1 the investigator remotely reviews the results of the V-2 exams and authorizes the performance of the V-1 radiological exams (MRI and Total-Body PET Scan) in the radiology center.

In the V0, the PI and his team perform the baseline UHDRS and body weight assessments. The patient will be randomized to Nestacell® or placebo. Those weighing 50 to 67.9 kg will receive 100 million cells (or placebo) and those weighing ≥ 68 kg will receive 136 million cells(or placebo) per administration. The doses are based on the V0 weight assessment and will not change throughout the study unless the PI asks for safety reasons (for example, a relevant weight loss).

The V1 marks the first investigational product administration. It will happen in sites unrelated to those performing the outcomes evaluation by personnel specially trained to prepare and administer the investigational product. After the females with childbearing potential performe the urine pregnancy test, NestaCell® or placebo will be administered intravenously in three cycles of three-monthly administrations with a monthly interval between cycles (total of 9 administrations). The other administrations happen at visits V2, V3, V5, V6, V7, V9, V10, and V11. To assure blindness, UHDRS and other clinical evaluations will be carried out in the research center [by the principal investigator (PI)] while the administrations will be made in the Center for the Investigational Product Administration (CIPA). The outcome evaluations by the PI and his/her team happen at V4, V8, and V12, one month after the end of each cycle. In the V13, the patients will also be directed to the radiology center to repeat the MRI exam.

Each patient participates in the trial for approximately 14 months, two months for screening, and twelve months for investigational product administration and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Age from 18 to 55 years;
3. HD diagnostic confidence level (DCL) score of 3 or 4 at enrolment;
4. HD manifestations begin from 4 to 8 years before enrolment;
5. UHDRS Total Functional Capacity (TFC) from 7 to 12, suggesting mild-moderate functional impairment;
6. Body weight at the V -1 from 50 to 90 Kg;
7. CAG repeats from 40 to 50;
8. ICF signature.

Exclusion Criteria:

1. Juvenile Huntington's disease,
2. Concomitant epilepsy;
3. Decompensated psychiatric disorders;
4. History of a suicide attempt;
5. Other neurological or musculoskeletal disorders that might interfere with the assessments;
6. Prior use of gene or cell therapy.
7. Confirmed or suspected cancer within the last 1 year (except operated basal cell carcinoma);
8. History of allergy to imaging exams contrast, or bovine origin products;
9. Current or planned use of immunosuppressants;
10. Clinically significant changes in the safety exams, defined as;

    * Serum transaminases (ALT, AST) increased > 2.5 × upper limit of normality (ULN).
    * Absolute neutrophil count in peripheral blood < 3,000 cells/1 mm3.
    * Serum creatinine > 2 × age- and sex-specific ULN.
    * Positive serology for HIV 1 and 2 (Anti-HIV-1,2), HTLV I and II, HBV (HBsAg, Anti-HBc), HCV (anti-HCV-Ab), and FTA-ABS.
    * Amylase, Troponin I, CKmB increased > 2.0 × ULN.
    * Malignancy shown by the Total-Body PET Scan.
    * Glycated hemoglobin > 6.5%.
    * aPTT, TT, platelets > 2.5 x ULN.
11. Pregnancy, lactation, or pregnancy plan;
12. BMI less than 18.5 at enrolment;
13. Participation in a clinical trial within twelve months before inclusion;
14. History of surgical procedures aiming at improving symptoms of Huntington's disease, such as neural transplantations, lesions of the central nervous system, infusions of neurotrophic agents, or deep brain stimulation.
15. Any medical condition that makes the patient unsuitable for the study or increases the risk of participation at the investigator's discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-08 (Estimated); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective | 1 year
  Proportion of patients who stabilized or decreased the UHDRS-TMS from Visit 0 to Visit 12 in the Nestacell® vs. Placebo groups.

SECONDARY OUTCOMES:
Secondary Efficacy Objectives | 1 year
  Mean variation of the UHDRS-TMS mean variation from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Proportion of patients who stabilized or increased the UHDRS-TFC from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Mean variation of the UHDRS-TFC from Visit 0 to Visit 12 of the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Proportion of patients who stabilized or increased the cUHDRS from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Mean variation of the cUHDRS from Visit 0 to Visit 12 of the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Proportion of patients who stabilized the MRI outcomes: 7.1 white substance, 7.2 gray substance, from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Mean variation of the MRI outcomes: 8.1 white substance, 8.2 gray substance, from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Proportion of patients who stabilized or decreased the NfL blood levels from Visit 0 to Visit 12 in the groups Nestacell® and Placebo.
Secondary Efficacy Objectives | 1 year
  Mean variation of the NfL blood levels from Visit 0 to Visit 12 of the groups Nestacell® and Placebo.

OTHER OUTCOMES:
Secondary Safety Objective | 1 year
  Occurrence, severity and cause of adverse events related to the study drug
Exploratory objectives | 1 year
  Blood concentration of nestin, IL-6, IL-17, TNFα, IFN-γ, C-reactive protein, BDNF, PT, aPTT, and D-dimer and the saliva concentration of BDNF and huntingtin before and 24 h after the NestaCell® administration at V1 and in a subset of 20-30 HD patients.
Exploratory objectives | Up to 9 months
  Blood concentration of nestin, IL-6, IL-17, TNFα, IFN-γ, C-reactive protein, BDNF, PT, aPTT, and D-dimer and the saliva concentration of BDNF and huntingtin before and 24 h after the NestaCell® administration at V9 in a subset of 20-30 HD patients.
Exploratory objectives | Up to 9 months
  Evolution between V1 and V9 of the blood concentration of nestin, IL-6, IL-17, TNFα, IFN-γ, C-reactive protein, BDNF, PT, aPTT, and D-dimer and the saliva concentration of BDNF and huntingtin before the NestaCell® administration in a subset of 20-30 HD patients
Exploratory objectives | Up to 9 months
  Evolution between V1 and V9 of the blood concentration of nestin, IL-6, IL-17, TNFα, IFN-γ, C-reactive protein, BDNF, PT, aPTT, and D-dimer and the saliva concentration of BDNF and huntingtin 24 hours after the NestaCell® administration in a subset of 20-30 HD patients.
Exploratory objectives | 1 year
  Measure of the relative amount of study participants who experienced changes in hair color during the course of the study.Nestacell® and placebo groups.
Exploratory objectives | 1 year
  Measure of the relative number of study participants who experienced hair growth.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Ferrara, Doctor, Study Director — Azidus Brasil

IPD SHARING:
Plan to Share IPD: No
After the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.

REFERENCES:
- [Background] ABH - Associação Brasil Huntington. p. Perguntas Frequentes. Disponível em: https://abh.org.br/perguntas-frequentes/. Acesso em: 19/12/2022.
- [Background] BARRETO, R. D. R. Características da Disfunção Congnitiva na Doença de Huntington. Orientador: JANUÁRIO, D. C. 2009. 87 f. (Mestre) - Faculdade de Medicina, Universidade de Coimbra.
- [Background] Bathina S, Das UN. Brain-derived neurotrophic factor and its clinical implications. Arch Med Sci. 2015 Dec 10;11(6):1164-78. doi: 10.5114/aoms.2015.56342. Epub 2015 Dec 11. PMID 26788077
- [Background] Baydyuk M, Xu B. BDNF signaling and survival of striatal neurons. Front Cell Neurosci. 2014 Aug 28;8:254. doi: 10.3389/fncel.2014.00254. eCollection 2014. PMID 25221473
- [Background] Benedict RH, DeLuca J, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the Symbol Digit Modalities Test as a cognition performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):721-733. doi: 10.1177/1352458517690821. Epub 2017 Feb 16. PMID 28206827
- [Background] BENTON, A. L.; HAMSHER, K. S.; SIVAN, A. B.; PSYCHOLOGICAL ASSESSMENT RESOURCES, I. Multilingual Aphasia Examination, Third Edition: Manual of instructions. PAR, 1978.
- [Background] Biglan KM, Zhang Y, Long JD, Geschwind M, Kang GA, Killoran A, Lu W, McCusker E, Mills JA, Raymond LA, Testa C, Wojcieszek J, Paulsen JS; PREDICT-HD Investigators of the Huntington Study Group. Refining the diagnosis of Huntington disease: the PREDICT-HD study. Front Aging Neurosci. 2013 Apr 2;5:12. doi: 10.3389/fnagi.2013.00012. eCollection 2013. PMID 23565093
- [Background] Chen J, Marks E, Lai B, Zhang Z, Duce JA, Lam LQ, Volitakis I, Bush AI, Hersch S, Fox JH. Iron accumulates in Huntington's disease neurons: protection by deferoxamine. PLoS One. 2013 Oct 11;8(10):e77023. doi: 10.1371/journal.pone.0077023. eCollection 2013. PMID 24146952
- [Background] Dorsey ER, Beck CA, Darwin K, Nichols P, Brocht AF, Biglan KM, Shoulson I; Huntington Study Group COHORT Investigators. Natural history of Huntington disease. JAMA Neurol. 2013 Dec;70(12):1520-30. doi: 10.1001/jamaneurol.2013.4408. PMID 24126537
- [Background] FDA. Guidance for Industry: Considerations for the Design of Early-Phase Clinical Trials of Cellular and Gene Therapy Products. pp. 27.
- [Background] Frank S, Testa C, Edmondson MC, Goldstein J, Kayson E, Leavitt BR, Oakes D, O'Neill C, Vaughan C, Whaley J, Gross N, Gordon MF, Savola JM; Huntington Study Group/ARC-HD Investigators and Coordinators. The Safety of Deutetrabenazine for Chorea in Huntington Disease: An Open-Label Extension Study. CNS Drugs. 2022 Nov;36(11):1207-1216. doi: 10.1007/s40263-022-00956-8. Epub 2022 Oct 15. PMID 36242718
- [Background] GAMARRA, L.; CINTRA, L.; GÁRATE, A. P. Relatório Final do Estudo de Biodistribuição do Produto NestaCell®. Centro de Experimentação e Treinamento em Cirurgia (CETEC) do Instituto Israelita de Ensino e Pesquisa Hospital Albert Einstein, p. 72. 2022.
- [Background] Unified Huntington's Disease Rating Scale: reliability and consistency. Huntington Study Group. Mov Disord. 1996 Mar;11(2):136-42. doi: 10.1002/mds.870110204. PMID 8684382
- [Background] JANUÁRIO, C. Doença de Huntington. Onde estamos agora? 2011. 148 f. (Doutor) -, Universidade de Coimbra.
- [Background] Muller M, Leavitt BR. Iron dysregulation in Huntington's disease. J Neurochem. 2014 Aug;130(3):328-50. doi: 10.1111/jnc.12739. Epub 2014 May 28. PMID 24717009
- [Background] Niu L, Ye C, Sun Y, Peng T, Yang S, Wang W, Li H. Mutant huntingtin induces iron overload via up-regulating IRP1 in Huntington's disease. Cell Biosci. 2018 Jul 4;8:41. doi: 10.1186/s13578-018-0239-x. eCollection 2018. PMID 30002810
- [Background] PATTERSON, J. Verbal Fluency. In: KREUTZER, J. S.;DELUCA, J., et al (Ed.). Encyclopedia of Clinical Neuropsychology. New York, NY: Springer New York, 2011. p. 2603-2606.
- [Background] Pringsheim T, Wiltshire K, Day L, Dykeman J, Steeves T, Jette N. The incidence and prevalence of Huntington's disease: a systematic review and meta-analysis. Mov Disord. 2012 Aug;27(9):1083-91. doi: 10.1002/mds.25075. Epub 2012 Jun 12. PMID 22692795
- [Background] Resolução CNS nº 466. Brasília: Conselho Nacional de Saúde 2012.
- [Background] Resolução RDC n°508. Brasilia: Conselho Nacional de Saúde 2021.
- [Background] SPREEN, O.; SPREEN, B. P. P. O.; STRAUSS, E.; STRAUSS, P. P. E. A Compendium of Neuropsychological Tests: Administration, Norms, and Commentary. Oxford University Press, USA, 1998. 9780195100198.
- [Background] Tumas V, Camargos ST, Jalali PS, Galesso Ade P, Marques W Jr. Internal consistency of a Brazilian version of the unified Huntington's disease rating scale. Arq Neuropsiquiatr. 2004 Dec;62(4):977-82. doi: 10.1590/S0004-282X2004000600009. Epub 2004 Dec 15. PMID 15608955
- [Background] Walker FO. Huntington's disease. Lancet. 2007 Jan 20;369(9557):218-28. doi: 10.1016/S0140-6736(07)60111-1. PMID 17240289
- [Background] Wenceslau CV, de Souza DM, Mambelli-Lisboa NC, Ynoue LH, Araldi RP, da Silva JM, Pagani E, Haddad MS, Kerkis I. Restoration of BDNF, DARPP32, and D2R Expression Following Intravenous Infusion of Human Immature Dental Pulp Stem Cells in Huntington's Disease 3-NP Rat Model. Cells. 2022 May 17;11(10):1664. doi: 10.3390/cells11101664. PMID 35626701